CLINICAL TRIAL: NCT02353572
Title: A Phase I-II Study of Infusional Melphalan + Bortezomib for Myeloablative Therapy Prior to Autologous Transplant for Patients With Multiple Myeloma
Brief Title: Melphalan and Bortezomib Prior to Autologous Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Principle investigator left the institution
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0817.cc
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-01

CONDITIONS: Plasma Cell Myeloma; Plasmacytosis; Recurrent Plasma Cell Myeloma; Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Melphalan; Bortezomib; Dexamethasone; Calcium Dobesilate; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melphalan, Bortezomib, Autologous transplant (Experimental): Patients receive melphalan IV continuously on days -5 to -2 and bortezomib IV over 3-5 seconds on days -4 and -1. Patients also receive dexamethasone IV on day -1 prior to the second dose of bortezomib. Beginning two days after completion of melphalan infusion, patients undergo autologous hematopoietic stem cell transplant. Eligible patients may undergo a second transplant 2-4 months after completion of the first transplant.
  Interventions: Drug: Melphalan; Drug: Bortezomib; Drug: Dexamethasone; Procedure: Autologous Transplant

INTERVENTIONS:
Drug: Melphalan — Given IV
  Other Names: Alkeran
Drug: Bortezomib — Given IV
  Other Names: Velcade
Drug: Dexamethasone — Given IV
  Other Names: Decadron, Ozurdex, Maxidex, Baycadron
Procedure: Autologous Transplant — Undergo autologous hematopoietic stem cell transplant
  Other Names: Autologous Hematopoietic Stem Cell Transplantation

SUMMARY:
This phase I/II trial studies the safety and best dose of melphalan and bortezomib when given prior to an autologous stem cell transplant and to see how well they work in treating patients with multiple myeloma. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bortezomib may help melphalan work better by making cancer cells more sensitive to the drug. Giving chemotherapy before an autologous hematopoietic stem cell transplant helps kill any cancer cells that are in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Giving melphalan together with bortezomib prior to autologous hematopoietic stem cell transplant may be a better treatment for multiple myeloma.

DETAILED DESCRIPTION:
This is a phase I, dose-escalation study of melphalan and bortezomib followed by a phase II study.

Patients receive melphalan intravenously (IV) continuously on days -5 to -2 and bortezomib IV over 3-5 seconds on days -4 and -1. Patients also receive dexamethasone IV on day -1 prior to the second dose of bortezomib. Beginning two days after completion of melphalan infusion, patients undergo autologous hematopoietic stem cell transplant. Eligible patients may undergo a second transplant 2-4 months after completion of the first transplant.

After completion of study treatment, patients are followed up monthly for at least 1 year and then every 3-6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic active multiple myeloma requiring treatment, including those whose prior smoldering myeloma progressed to symptomatic disease requiring chemotherapy; both newly diagnosed and previously treated patients are eligible for the study
* Presence of quantifiable M-component of immunoglobulin G (IgG), IgA, IgD, or IgE and/or urinary kappa or lambda light chain or Bence Jones protein, in order to evaluate response; non-secretory patients are eligible provided the patient has > 20% plasmacytosis or multiple (> 3) focal plasmacytomas on magnetic resonance imaging (MRI) or diffuse hyperintense signal on short tau inversion recovery (STIR) weighted images
* Performance status of 0-2 based on Southwest Oncology Group (SWOG) criteria; patients with a poor performance status (3-4) are also eligible after having improved their performance to 0-2
* No significant co-morbid medical conditions; no uncontrolled life threatening infection
* Patient evaluation should be done within 35 days prior to registration; signed informed consent should be obtained from all patients in accordance with institutional and federal guidelines

Exclusion Criteria:

* Patients with a history of recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, difficult to control significant cardiac arrhythmias, or arrhythmia associated with prolonged QT interval; left ventricular ejection fraction by echocardiogram or multi gated acquisition scan (MUGA) < 45% assessed within 35 days prior to study registration
* Patients with a history of moderate to severe chronic obstructive and/or restrictive pulmonary disease, with a forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) < 50% of the predicted values; diffusing capacity of the lung for carbon monoxide (DLCO) < 50%; partial pressure of oxygen (P02) < 70 mmHg
* Patients with a prior history of malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years
* Pregnant or nursing women; women of child-bearing potential must have a negative pregnancy documented within one week of registration; women/men of reproductive potential may not participate unless they have agreed to use two forms of effective contraceptive method
* Human immunodeficiency virus (HIV) positive patients
* Transaminases > 2 x normal values or bilirubin > 2 x normal values; prior history of chronic liver disease
* Patients with renal failure on dialysis
* Active uncontrolled infection
* History of significant psychiatric illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Choon-Kee Lee, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2009 and September 2011, 3 patients were enrolled in the study from University of Colorado Cancer Center
Pre-assignment Details: Within 35 days of planned therapy, patients were evaluated for eligibility by standard tests: paraprotein assessment, bone marrow biopsy and aspiration, MRI scan, PET/CT scan, echocardiography and pulmonary function test. Patients who were not be able to pursue the tandem autotransplant were eligible for one autotransplant.
Groups:
- Melphalan, Bortezomib, Autologous Transplant: Patients received melphalan IV continuously on days -5 to -2 and bortezomib IV over 3-5 seconds on days -4 and -1. Patients also received dexamethasone IV on day -1 prior to the second dose of bortezomib. Beginning two days after completion of melphalan infusion, patients underwent autologous hematopoietic stem cell transplant.
Period: Overall Study
Arm/Group | Melphalan, Bortezomib, Autologous Transplant
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Study terminated | 2

BASELINE CHARACTERISTICS:
Population: Based on the annual number of referrals made to the Myeloma and Amyloidosis Program, expected accrual to this study was about 20 patients per year.
Arm/Group | Melphalan, Bortezomib, Autologous Transplant
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerable Dose (MTD) of Both Melphalan and Bortezomib as Combination
Description: MTD is defined as one dose below that which 33% of patients within cohort experienced dose limiting toxicity. Unacceptable toxicity is defined as intractable veno-occlusive disorder, new onset of renal failure requiring dialysis, acute heart failure of New York Heart Association class III/IV, or interstitial pneumonia requiring ventilator management for longer than 3 days or grade 4 neuropathy. A 100-day mortality/toxicity rate of 3% or more is considered unacceptable. Will consider as evidence an observed 100-day mortality/toxicity rate whose lower one-sided 90% confidence bound exceeds 3%.
Time Frame: 100 days
Population: The study was terminated, study endpoints were not reached.
Arm/Group | Melphalan, Bortezomib, Autologous Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events for approximately 1 year until the study was terminated.
Arm/Group | Melphalan, Bortezomib, Autologous Transplant
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
This study was terminated due to the investigator's departure from the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes